CLINICAL TRIAL: NCT04529785
Title: Added Value of Vein of Marshal Ethanol Infusion Compared to Superior Vena Cava Isolation Alone in Patients Undergoing Repeat Ablation for Recurrent Paroxysmal Atrial Fibrillation Despite Durable Pulmonary Vein Isolation
Brief Title: Added Value of Vein of Marshal Ethanol Infusion Compared to Superior Vena Cava Isolation Alone in Patients Undergoing Repeat Ablation for Recurrent Paroxysmal Atrial Fibrillation Despite Durable PV Isolation
Acronym: VEIN-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Sebastien Knecht, Professor Doctor, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2700
Record Dates: First submitted 2020-08-20; First posted 2020-08-28 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SVC only (Active Comparator): Patients in Group 1 will receive an SVC isolation only
  Interventions: Procedure: SVC only
- SVC isolation with substrate modification and VoM inf (Active Comparator): Patients in Group 2 will receive an SVC isolation with substrate modification and vein of Marshal ethanol infusion
  Interventions: Procedure: SVC isolation with substrate modification and vein of Marshal ethanol infusion

INTERVENTIONS:
Procedure: SVC only — Patients allocated to this arm will receive an RF ablation with the isolation of the SVC alone
  Arms: SVC only
Procedure: SVC isolation with substrate modification and vein of Marshal ethanol infusion — Patients allocated to this arm will receive an RF ablation with the isolation of the SVC, substrate modification and vein of Marshal ethanol infusion
  Arms: SVC isolation with substrate modification and VoM inf

SUMMARY:
The superior vena cava (SVC) is one of the most common non pulmonary vein (PV)-triggers for atrial tachyarrhythmias. SVC electrical isolation can be reached by circular radiofrequency (RF)-ablation under close monitoring of the phrenic nerve. However, adding substrate modification and vein of Marshal (VoM) ethanol infusion to the ablation procedure might substantially improve long-term outcomes.

The aim of this study is to evaluate the recurrence rate 1 year after the index ablation in patients undergoing a redo ablation for recurrent paroxysmal atrial fibrillation (PAF) despite durable pulmonary vein isolation (PVI) with either SVC isolation alone or with substrate modification including vein of Marshal ethanolisation in addition to SVC isolation alone

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients scheduled for a repeat ablation of PAF after a previous PVI
* Confirmation of lasting pulmonary vein isolation at the time of randomization

Exclusion Criteria:

* Patients with persistent atrial fibrillation
* Previous ablation with isolation of the SVC, roofline, mitral line or previous vein of Marshal ethanol infusion
* Left atrial thrombus. Left atrial appendage thrombus can be determined by preprocedural imaging: CT, transesophageal echocardiography or MRI.
* Left ventricular ejection fraction <35%.
* Cardiac surgery within the previous 90 days.
* Expecting cardiac transplantation or other cardiac surgery within 180 days.
* Coronary percutaneous transluminal coronary angioplasty/stenting within the previous 90 days or myocardial infarction within the previous 60 days.
* Documented history of a thromboembolic event within the previous 90 days.
* Diagnosed atrial myxoma.
* Significant restrictive, constrictive, or chronic obstructive pulmonary disease with chronic symptoms.
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment
* Women who are pregnant or who plan to become pregnant during the study.
* Acute illness or active infection at time of index procedure
* Advanced renal insufficiency
* Unstable angina.
* History of blood clotting or bleeding abnormalities.
* Contraindication to anticoagulation.
* Life expectancy less than 1 year.
* Presence of a condition that precludes vascular access.
* International Normalized Ratio greater than 3.5 within 24 hours of procedure - for patients taking warfarin.
* Patient cannot be removed from antiarrhythmic drugs for reasons other than AF.
* Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial tachyarrhythmia 1 year after the index ablation | 1 year
  Comparison of the prevalence of atrial tachyarrhythmia recurrence 1 year after the index ablation between groups
Safety (complications) | During procedure
  Comparison of the number of procedural complications between groups

SECONDARY OUTCOMES:
Total procedural time | During procedure
  Comparison of the procedural time between groups
Fluoroscopy time | During procedure
  Comparison of the fluoroscopy time between groups
RF ablation time | During procedure
  Comparison of the radiofrequency time between groups

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Knecht, MD, PhD, Principal Investigator — AZ Sint-Jan AV
Locations (1):
- AZ Sint-Jan Brugge-Oostende AV, Bruges, Please Select, Belgium

IPD SHARING:
Plan to Share IPD: No